CLINICAL TRIAL: NCT05538338
Title: Intrauterine Platelet Rich Plasma (PRP) Infusion for Endometrial Insufficiency: A Prospective, Double-Blind, Placebo-Controlled Randomized Controlled Trial
Brief Title: Platelet Rich Plasma for Insufficient Endometrium
Acronym: PIER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RMA-2022-04
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Infertility of Uterine Origin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): an intrauterine infusion of platelet rich plasma (PRP) will be administered to this group
  Interventions: Other: Platelet Rich Plasma Intrauterine infusion
- Control Group (Placebo Comparator): an intrauterine infusion of normal saline will be administered to this group
  Interventions: Other: Normal saline Intrauterine infusion

INTERVENTIONS:
Other: Platelet Rich Plasma Intrauterine infusion — an intrauterine infusion of platelet rich plasma (PRP) will be administered to this group of participants
  Arms: Intervention Group
Other: Normal saline Intrauterine infusion — an intrauterine infusion of normal saline will be administered to this group of participants
  Arms: Control Group

SUMMARY:
To determine the effectiveness of an intrauterine PRP infusion on endometrial thickness and in vitro fertilization (IVF) outcomes in a population of infertile women with a history of unresponsive thin endometrium.

DETAILED DESCRIPTION:
Patients with a history of thin endometrium will be randomized to either an intrauterine infusion of PRP vs. a placebo infusion of normal saline. This is a double-blind, placebo controlled prospective RCT. Patients will then proceed with a frozen embryo transfer of a single euploid embryo per routine.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have previously undergone at least 2 unsuccessful frozen embryo transfer cycles, defined as failure to achieve a sustained clinical pregnancy (visualization of intrauterine gestational sac on ultrasound or a cancelled embryo transfer cycle due to inadequate endometrial thickness
* Patients with a diagnosis of thin endometrial lining (less than or equal to 6 mm maximum thickness) during prior unsuccessful or canceled embryo transfer cycles.

Exclusion Criteria:

* Fewer than 2 prior unsuccessful or canceled frozen embryo transfer cycles.
* Most recent unsuccessful embryo transfer prior to January 1, 2017.
* Mullerian anomalies, excluding arcuate uterus
* Concurrent submucosal fibroids, unrepaired uterine defects or present indication for uterine surgery
* Communicating hydrosalpinx without plans for surgical correction prior to study enrollment.
* Failure of patient to agree to enrollment in study with written consent.
* Concurrent pregnancy
* Anticoagulation use for which plasma infusion is contraindicated
* History of thrombosis
* Thrombophilia either inherited or acquired
* Concomitant use of adjunctive therapies for proliferation. These must be discontinued upon enrollment.
* Embryo planned to be used for transfer generated from surgically obtained sperm due to a diagnosis of non-obstructive azoospermia
* Recurrent/persistent endometrial fluid in prior cycles

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Endometrial Thickness during frozen embryo transfer | during the proliferative phase of the frozen embryo transfer cycle
  peak endometrial thickness prior to initiation of progesterone

SECONDARY OUTCOMES:
Sustained implantation rate | approximately 9 weeks gestational age
  presence of fetal heart beat upon discharge from care

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No